CLINICAL TRIAL: NCT05161104
Title: A Multicenter Cross-sectional Study of Cardiac Ultrasound Phenotypes in Patients With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiuling Shang, Clinical Professor, Fujian Provincial Hospital
Other Study IDs: K2021-10-001
Record Dates: First submitted 2021-11-23; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Ultrasound Phenotypes; Septic Myocardial Suppression; Hyperdynamic State Left Ventricular Function in Sepsis Patients; Outcome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- left ventricular systolic dysfunction(LVSD)
- left ventricular diastolic dysfunction(LVDD)
- right ventricular dysfunction(RVD)
- diffuse ventricular dysfunction
- hyperdynamic state left ventricular function
- Normal

SUMMARY:
The heart, one of the most important organs for oxygen supply and consumption, is frequently involved in sepsis, i.e. septic cardiomyopathy, also known as septic myocardial suppression. The occurrence of septic myocardial suppression increases mortality in septic patients. Recent studies have found that left ventricular hyperdynamic state (EF > 70%) is associated with intra-ICU mortality in septic patients, possibly because it reflects unresolved vascular paralysis from sepsis . For septic myocardial suppression, there is still a lack of uniform criteria for diagnosis, but it is well established that the cardiac ultrasound phenotype of septic myocardial suppression can be left ventricular systolic insufficiency (LVSD), left ventricular diastolic insufficiency (LVDD), right ventricular insufficiency (RVD), diffuse ventricular insufficiency, and mixed ventricular insufficiency. According to incomplete statistics, the prevalence of LVSD ranges from 12 to 60%, the prevalence of LVDD is higher, 20% to 79%, and the prevalence of RVD varies from 30% to 55%. However, based on the current understanding of septic myocardial suppression, the relationship between each staging and its prognosis is unclear, and echocardiography can rapidly identify septic myocardial suppression and guide the classification of septic myocardial suppression to further optimize the diagnosis and treatment process of sepsis, especially to avoid over-resuscitation during fluid resuscitation and perform reverse resuscitation in a timely manner to improve patient prognosis and reduce hospitalization time. The aim of this study is to classify and evaluate the prognosis of patients with different septic cardiac ultrasound phenotypes in multiple centers across China by measuring the right and left heart systolic and diastolic indices by echocardiography, recording the baseline conditions and clinical indices of patients, and combining them with the prognosis.

ELIGIBILITY:
Inclusion Criteria:

- All patients with sepsis or septic shock who conform to Sepsis 3.0 diagnostic criteria

Exclusion Criteria:

1. Patients with preexisting chronic heart disease such as cardiomyopathy, chronic pulmonary heart disease, severe cardiac valve disease, coronary heart disease, congenital heart disease, pericardial disease, etc. and with cardiac function ≥ grade III (NYHA classification) prior to sepsis.
2. End-stage malignancies.
3. Severe trauma.
4. Pregnancy.
5. Patients for whom transthoracic echocardiography data are not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with sepsis or septic shock who conform to Sepsis 3.0 diagnostic criteria and were more than or equal to 18 years of age who were admitted to each center were included. Sepsis was defined as an increase of ≥2 points from baseline in sequential organ failure assessment (SOFA) score due to infection; septic shock was defined as persistent hypotension on top of sepsis, requiring vasoactive drugs to maintain a mean arterial pressure(MAP) ≥65 mmHg and a blood lactate level >2 mmol/L despite adequate fluid resuscitation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-11-23 (Estimated); Study Completion 2025-11-23 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Number of patient deaths divided by the total number
28-day mortality | From patient admission to day 28
  Number of patient deaths within 28 days divided by the total number

SECONDARY OUTCOMES:
length of stay in the ICU | days from patient transfer to ICU to transfer out，an average of 1 week
  Total number of days from patient transfer to ICU to transfer out of ICU
number of days of mechanical ventilation | Days the patient was mechanically ventilated until the cessation of mechanical ventilation，an average of 1 week
  Total number of days the patient was mechanically ventilated until the cessation of mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Zhang H, Wang X, Yin W, Zhang H, Liu L, Pan P, Zhu Y, Huang W, Xing Z, Yao B, Wang C, Lin T, Yu R, Shang X. A multicenter prospective cohort study of cardiac ultrasound phenotypes in patients with sepsis: Study protocol for a multicenter prospective cohort trial. Front Med (Lausanne). 2022 Jul 27;9:938536. doi: 10.3389/fmed.2022.938536. eCollection 2022. PMID 35966841